CLINICAL TRIAL: NCT05740501
Title: Pharmacokinetic Profiling of Pembrolizumab (Keytruda&Amp;Reg;) and Nivolumab (Opdiva&Amp;Reg;) in Patients With Melanoma and/or Non-Small Cell Lung Cancer: Clinical Validation of a Mass Spectrometry-based Assay
Brief Title: Pharmacokinetic Profiling of Pembrolizumab and Nivolumab in Patients With Melanoma and/or Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Paul Jannetto, Principal Investigator, Mayo Clinic
Other Study IDs: 17-002103; NCI-2023-00069 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-02-03; First posted 2023-02-23 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Lung Non-Small Cell Carcinoma; Melanoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection, chart review): Patients undergo collection of blood samples and have medical records reviewed on study.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Medical records are reviewed
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This early phase I study collects blood samples and monitors the levels of pembrolizumab and nivolumab as they move through the body in patients with melanoma and/or non-small cell lung cancer. Pembrolizumab and nivolumab are a monoclonal antibodies that may interfere with the ability of cancer cells to grow and spread. Studying samples of blood in the laboratory from patients receiving pembrolizumab and nivolumab may help doctors learn more about the effects of pembrolizumab and nivolumab on cells. It may also help doctors understand how well patients respond to treatment. Information from this study may be used in the future to guide physicians to make dosage adjustments based on serum concentrations of drug to minimize adverse side effects and maximize the effect of the drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To perform a steady-state PK study on patients who are taking monoclonal antibody therapy (25 patients starting pembrolizumab and 25 patients starting nivolumab for melanoma or non-small cell lung cancer).

II. Develop and validate a liquid chromatography tandem mass spectrometry (LC-MS/MS) assay to measure pembrolizumab and nivolumab in serum.

III. Measure patient samples for pembrolizumab/nivolumab at various clinical time points.

IV. Use the pharmacokinetic data (drug concentrations) to determine the area under the curve (AUC), maximum observed serum concentration (Cmax), clearance, half-life (t1/2), and trough steady-state drug concentrations.

V. Compare the data to the clinical efficacy (defined using Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria)1, as well as, presence of auto-immune side effects using multiple variable regression modeling in Statistical Analysis System (SAS) version (v)9.4 or other statistical software.

OUTLINE:

Patients undergo collection of blood samples and have medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are at steady-state and taking monoclonal antibody therapy with pembrolizumab or nivolumab for melanoma or non-small cell lung cancer. Steady-state for pembrolizumab is week 21 or later and for nivolumab is week 14 or later from the initial infusion

Exclusion Criteria:

* Patients not taking pembrolizumab or nivolumab or taking pembrolizumab or nivolumab for other indications (not melanoma or non-small cell lung cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with melanoma or non-small cell lung cancer who are taking monoclonal antibody therapy at Mayo Clinic Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Development and validation of a laboratory developed test (LDT) using liquid chromatography tandem mass spectrometry to measure pemborlizumab and nivolumab. | Up to 1 year
  Verify the accuracy, precision, linearity, sensitivity and specificity of a mass spectrometry assay for pembrolizumab and nivolumab in serum
Measurement of patient samples for pembrolizumab | Through study completion at several time points, an average of 3 weeks after taking pembrolizumab for at least 21 weeks.
  Using a validated LDT liquid chromatography tandem mass spectrometry assay measure the concentration of pembrolizumab in serum.
Measurement of patient samples for nivolumab | Through study completion at several time points, an average of 1 month after taking nivolumab for at least 14 weeks
  Using a validated LDT liquid chromatography tandem mass spectrometry assay measure the concentration of nivolumab in serum.
Correlation of steady-state concentrations of pembrolizumab correlate with clinical efficacy and/or toxicity | Through study completion, an average of 3 weeks after taking pembrolizumab for at least 21 weeks.
  Will assess if therapeutic drug monitoring correlates with efficacy and/or toxicity of pembrolizumab. Concentrations in serum will be determined using a LDT mass spectrometry assay.
Correlation of steady-state concentrations of nivolumab correlate with clinical efficacy | Through study completion, an average of 1 month after taking nivolumab for at least 14 weeks
  Will assess if therapeutic drug monitoring correlates with efficacy and/or toxicity of nivolumab. Concentrations in serum will be determined using a LDT mass spectrometry assay.
Clinical efficacy | After 6 months (24 weeks or more) of treatment
  Tumor response will be determined using Response Evaluation Criteria in Solid Tumors1.1 criteria. Clinical efficacy defined as achieving an objective response (complete response or partial response) versus stable disease, or disease progression.
Presence of auto-immune side effects | Through study completion, an average of 1 month
  Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse events, version 4.0. Investigators will indicate if it was potentially immune related (i.e. grade 3-4 adverse events such as pneumonitis, diarrhea/colitis, hypophysitis/adrenal insufficiency, hyper/hypothyroidism, autoimmune hepatitis, severe skin reactions, nephritis/kidney failure, uveitis, myositis) in combination with other basic laboratory tests that are routinely monitored. Will use multiple variable regression modeling in Statistical Analysis System version 9.4 or other statistical software.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Jannetto, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States